CLINICAL TRIAL: NCT05458427
Title: Dedicated Breast CT for Diagnosis of Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Unethical to include many more patients when currently obtained results are sufficient.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL55378.091.15
Record Dates: First submitted 2022-07-06; First posted 2022-07-14 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Computed Tomography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dedicated breast computed tomography (BCT) is being developed as a new x-ray based tomographic breast imaging method for early breast cancer detection and/or diagnosis. BCT results in isotropic high spatial resolution three-dimensional (3D) images coupled with high contrast resolution. It is hypothesized that BCT imaging used as a replacement of the additional mammographic views during diagnostic work-up will improve the accuracy of clinical standard diagnostic work-up.

DETAILED DESCRIPTION:
Rationale:

Dedicated breast computed tomography (BCT) is being developed as a new x-ray based tomographic breast imaging method for early breast cancer detection and/or diagnosis. BCT results in isotropic high spatial resolution three-dimensional (3D) images coupled with high contrast resolution. It is hypothesized that BCT imaging used as a replacement of the additional mammographic views during diagnostic work-up will improve the accuracy of clinical standard diagnostic work-up.

Objective:

The primary objective of this research project is to determine the improvement in the area under the receiver operating characteristics (ROC) curve of BCT for diagnosis of breast cancer compared to that of the standard diagnostic work-up. As secondary objectives, this analysis will be performed by lesion type (microcalcifications vs. soft tissue lesions).

Study design:

Single arm study with each subject being its own control

ELIGIBILITY:
Inclusion Criteria:

* Women age 50 or older

Initial schema:

- Women who are scheduled to undergo a diagnostic work-up following an abnormal screening mammogram with the suspicious finding NOT located in the axillary tail of the breast This initial inclusion criterion will be used until 85 subjects that result in a Breast Imaging Reporting and Data System (BI-RADS) 1 or 2 after clinical diagnostic work-up are recruited and imaged.

Subsequent schema:

- Women who underwent diagnostic work-up following an abnormal screening mammogram and were assigned a BI-RADS 4 or 5 due to soft tissue lesions (total 120 patients when combined with those from the initial schema), or due to microcalcifications (total 120 patients when combined with those from the initial schema) with the suspicious finding NOT located in the axillary tail of the breast

Each patient can only enroll once in the study.

Exclusion Criteria:

* Women who do not meet the inclusion criteria as described above
* Women with suspected or confirmed pregnancy
* Women who have had bilateral mastectomy
* Women whose suspicious lesion is located in the axillary tail
* Women with prior breast cancer or breast biopsy in the recalled breast in the last 12 months
* Women who are breastfeeding
* Women who are very frail and unable to cooperate
* Women who cannot give informed consent
* Male subjects

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population base consists of women recalled to undergo diagnostic work-up due to a suspicious finding at mammographic screening for breast cancer.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Probability of malignancy (POM) | One year after the end of participation in this study
  The primary objective of this study is to perform a prospective clinical trial to compare the performance of BCT and US (for soft tissue lesions) to that of the standard diagnostic work-up (several mammographic views and US for soft tissue lesions) for the diagnosis of breast cancer. The endpoint is the area under the receiver operating characteristic (ROC) curve (AUC) computed from probability of malignancy (POM) resulting from independent interpretation of the clinical diagnostic work-up images and the BCT images as produced by the BCT system + US (when acquired during standard clinical diagnostic workup).

SECONDARY OUTCOMES:
Probability of malignancy (POM) | One year after the end of participation in this study
  The secondary objective, a comparison is made among the clinical diagnostic work-up, the BCT images as produced by the system alone, and the BCT images enhanced using our novel algorithms alone. The endpoint is the area under the receiver operating characteristic (ROC) curve (AUC) computed from probability of malignancy (POM) resulting from independent interpretation images.

OTHER OUTCOMES:
Participant characteristics | Day of participation
  Participant characteristics such as age, gender, ethnicity, race, cup size, reason of referral, family history for breast cancer, level of comfort during BCT examination and level of comfort of BCT compared to other image modality.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Netherlands Cancer Institute, Amsterdam